CLINICAL TRIAL: NCT02990481
Title: A Phase 1, Multicenter, Open-label, Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of TRK-950 Given Intravenously in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study Evaluating the Safety of TRK-950 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 950P1V01
Record Dates: First submitted 2016-11-29; First posted 2016-12-13 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced or Metastatic Solid Carcinomas; Colon Cancer; Cholangiocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 - TRK-950 (Experimental): * Solid tumor
  * TRK-950 (Three dose levels will be explored during Arm 1)
  Interventions: Biological: TRK-950
- Arm 2 - TRK-950 (Experimental): * Colon cancer
  * TRK-950 (Low dose and High dose)
  Interventions: Biological: TRK-950
- Arm 3 -TRK-950 (Experimental): * Cholangiocarcinomas
  * TRK-950 (Low dose)
  Interventions: Biological: TRK-950

INTERVENTIONS:
Biological: TRK-950 — Intravenously over 60 minutes, on day 1, 8 and 15 of each cycle
  Arms: Arm 1 - TRK-950
Biological: TRK-950 — Low dose: intravenously over 60 minutes, on day 1, 8, 15 and 22 of each cycle
  High dose: intravenously over 60 minutes, on day 1 and 15 of each cycle
  Arms: Arm 2 - TRK-950
Biological: TRK-950 — Low dose: Intravenously over 60 minutes, on day 1, 8, 15 and 22 of each cycle
  Arms: Arm 3 -TRK-950

SUMMARY:
1. To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLTs) of TRK-950 as single agent
2. To establish the dose of TRK-950 recommended for future phase 2 studies

DETAILED DESCRIPTION:
This study is a first-in-human study of TRK-950 in patients with advanced solid tumors and is primarily designed to determine the dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of TRK-950 administered via intravenous (IV) infusion once weekly for 3 weeks every 28 days in Arm 1.

Once enrollment in Arm 1 was completed, two dose schedules will be evaluated in Arm 2 to determine the dosing schedule. Up to six (6) patients will be enrolled respectively.

In parallel, to determine anti-tumor activity up to twelve (12) patients will be enrolled in Arm 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed locally advanced or metastatic solid carcinomas in Arm 1
* Patients with histologically confirmed locally advanced or metastatic colon cancer in Arm 2
* Patients with histologically confirmed locally advanced or metastatic cholangiocarcinomas in Arm 3
* Tumor progression after receiving standard/approved chemotherapy or where there is no approved therapy or not amendable to a curative treatment
* Measurable disease per RECIST 1.1 (primary or metastases)

Exclusion Criteria:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or nursing women
* Treatment with radiation therapy, surgery, chemotherapy, immunotherapy, or investigational therapy within four weeks prior to study entry
* Unwillingness or inability to comply with procedures required in this protocol
* Known active infection with HIV, hepatitis B, hepatitis C
* Symptomatic brain metastases
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Adverse event | through study completion, an average of 1 year
CTCAE version 4.03 | through study completion, an average of 1 year
Blood pressure (mmHg) | through study completion, an average of 1 year
Heart rate (bpm) | through study completion, an average of 1 year
Respiratory rate (bpm) | through study completion, an average of 1 year
Temperature (°F or °C) | through study completion, an average of 1 year
Weight (lbs/kg) | through study completion, an average of 1 year
Height (inches/cm) | through study completion, an average of 1 year
Karnofsky performance status | through study completion, an average of 1 year
Electrocardiogram | through study completion, an average of 1 year
Clinical laboratory tests | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Area under the concentration curve(AUC) | through study completion, an average of 1 year
Maximum plasma concentration(Cmax) | through study completion, an average of 1 year
Time to maximum plasma concentration(Tmax) | through study completion, an average of 1 year
Terminal elimination half life(t1/2) | through study completion, an average of 1 year
Total body clearance(CL) | through study completion, an average of 1 year
Apparent volume of distribution(Vd) | through study completion, an average of 1 year
Tumor response rate | through study completion, an average of 1 year
Duration of response | through study completion, an average of 1 year
Time to progression | through study completion, an average of 1 year
Progression free survival | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okano F, Saito T, Minamida Y, Kobayashi S, Ido T, Miyauchi Y, Wasai U, Akazawa D, Kume M, Ishibashi M, Jiang K, Aicher A, Heeschen C, Yonehara T. Identification of Membrane-expressed CAPRIN-1 as a Novel and Universal Cancer Target, and Generation of a Therapeutic Anti-CAPRIN-1 Antibody TRK-950. Cancer Res Commun. 2023 Apr 18;3(4):640-658. doi: 10.1158/2767-9764.CRC-22-0310. eCollection 2023 Apr. PMID 37082579